CLINICAL TRIAL: NCT02346097
Title: ElectroCRT - Left Ventricular Lead Implant and Optimization Guided by Electrocardiography in Cardiac Resynchronization Therapy
Brief Title: Electrophysiological Optimization of Left Ventricular Lead Placement in CRT
Acronym: ElectroCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Electro-1-CRT
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Congestive Heart Failure
Keywords: Cardiac Resynchronization Therapy; Heart Failure; Ejection Fraction; Narrow; Pacemaker; Electrophysiology; Electrical activation mapping; Coronary Sinus; Mapping; QRS; QRS width; Pacing Interval; Left Ventricular Lead; Cardiac CT; Echocardiography; Myocardial Scintigraphy; 6 Minutes Walk Test; Imaging; Left ventricular ejection fraction; Epicardial veins; Resynchronization; ImagingCRT; Optimal electrical resynchronization; Cardiac computed tomography
MeSH Terms: conditions — Heart Failure; Aortic Coarctation | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal electrical resynchronization (Experimental): Cardiac Resynchronization Therapy: LV lead implant according to electrical activation mapping of available epicardial veins to identify the latest electrical activated myocardial region. Post-implant interventricular (VV) electrical optimization for narrowing the paced QRS width. Post-implant standard pacemaker settings: Atrioventricular (AV) interval 100-130 ms and VV interval settings with simultaneous biventricular pacing.
  Day 1 after implantation: ECG, AV-optimization guided by echocardiography, high-pitch cardiac CT to verify LV lead position.
  Programming of the VV interval to obtain the narrowest QRS-width
  Interventions: Device: Cardiac Resynchronization Therapy (St. Jude Qaudripolar LV lead)
- Routine CRT-strategy, imaging guided (Active Comparator): Cardiac Resynchronization Therapy: LV lead implant guided by echocardiography and Rb-PET towards the latest mechanically activated myocardial segment and separate from scar. Post-implant VV electrical optimization for narrowing the paced QRS width. Standard pacemaker settings for both groups: AV-interval 100-130 ms and VV-interval settings with simultaneous biventricular pacing.
  Day 1 after implantation: ECG, AV-optimization guided by echocardiography, high-pitch cardiac CT to verify LV lead position.
  Continue standard interventricular pacing interval settings with simultaneous pacing in both ventricular leads.
  Interventions: Device: Cardiac Resynchronization Therapy (St. Jude Qaudripolar LV lead)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (St. Jude Qaudripolar LV lead) — Optimal electrical resynchronization vs. routine CRT strategy, imaging guided. For more details refer to ""Arm descriptions"
  Other Names: St. Jude Qaudripolar LV lead

SUMMARY:
The purpose of this study is to investigate if "optimal electrical resynchronization" achieved by targeting left ventricular lead placement to the myocardial region with the latest electrical activation combined with post-implant pacemakersettings for narrowing the paced QRS width causes an excess improvement in the pumping function of the heart (the left ventricular ejection fraction) in Cardiac Resynchronization Therapy (CRT)

DETAILED DESCRIPTION:
Background:

Cardiac resynchronization therapy (CRT) is an established therapy in patients with a left ventricular (LV) ejection fraction (EF) < 35 %, and an electrocardiogram (ECG) with prolonged QRS duration (1). The treatment is implemented by implanting a pacemaker with three pacing leads: One in the right atrium, one in the right ventricle (RV) and one in an epicardial vein through the coronary sinus, thereby establishing atrial-synchronized biventricular pacing to coordinate RV and LV contraction.

Despite the convincing effect of CRT on survival, symptoms, and LV function (2,3,4) as much as 30-40 % of the patients do not benefit clinically from the treatment, so-called non-responders (5,6). Annually around 600 CRT-systems are implanted in Denmark and about 3000 patients live with a CRT. The risk of complications associated with CRT-treatment is considerable (7), and a conservative estimate of the expenses for implanting a CRT-device is DKK 80.000. Consequently, the costs of CRT in non-responders are high, both for the patients and for the health economy.

Potential correctable reasons for non-response to CRT are non-optimal LV lead positioning and non-optimal pacemaker programming (5). At the Department of Cardiology, Aarhus University Hospital, Skejby, the clinical practice is to place the LV lead in the non-apical postero-lateral region aiming towards a myocardial segment with electrical activation occurring in the second half of the QRS complex in the surface ECG.

Retrospective studies have documented an improved response rate to CRT when the LV lead is placed in a myocardial region with late electrical activation and without scar tissue (8,9). Furthermore, lack of electrical resynchronization after CRT illustrated by unchanged or prolonged QRS duration is associated with poor clinical outcome (10) and programming the interventricular (VV) delay to obtain the narrowest QRS-complex has been suggested to increase CRT response rate (11,12).

A recent randomized controlled trial (ImagingCRT) conducted at our institution demonstrated that an imaging guided LV lead placement strategy targeting the latest mechanically activated myocardial segment (assessed by pre-implant echocardiography) and separate from scar tissue (determined by pre-implant myocardial scintigraphy) improves clinical response rate to CRT (data not yet published). This method has the potential to become routine clinical practice for LV lead placement at our institution.

Aim and hypothesis:

We aim to investigate if optimal electrical resynchronization achieved by targeting LV lead placement to the myocardial region with the latest electrical activation determined by systematic electrical mapping of all available epicardial veins combined with post-implant VV electrical optimization for narrowing the paced QRS width causes an excess improvement in LVEF after CRT.

We hypothesize that this will cause an excess increase in LVEF of 4 %, to an absolute increase in LVEF of 12 % as compared to an absolute increase in LVEF to 8 % using an imaging guided CRT-implantation strategy.

Methods:

All patients referred to CRT at Aarhus University Hospital, Skejby will be assessed for eligibility. Eligibility criteria and outcomes measures elsewhere at clinicaltrial.gov.

Study Course:

After written informed consent the patient will follow the study course as specified below.

The day before implantation of the CRT the following investigations are scheduled: Echocardiography (to asses LV function and dimensions), cardiac CT-scan (to localize all available epicardial veins), myocardial scintigraphy (82Rubidium positron emission tomography (Rb-PET)), to determine the extent and distribution of scar tissue and LVEF (13,14)), blood samples and clinical evaluation.

The patients are randomized to EITHER imgaging guided placement of the LV lead targeting the myocardial region with the latest mechanical activation and VV-interval settings programmed with simultaneous biventricular pacing (routine CRT-strategy arm) OR LV lead placement guided by procedural electrical mapping of all available cardiac veins targeting the myocardial region with the latest electrical activation combined with VV electrical optimization the day after implantation to achieve the narrowest paced QRS width (intervention arm).

The day after the implantation all patients undergo a high-pitch cardiac CT to verify LV lead position (15), pacemaker test, programming of VV-intervals and echocardiographic atrioventricular (AV) optimization.

One month after the implantation all patients have their pacemaker tested by a research nurse according to standard clinical practice.

Six months after CRT implantation the following investigations are repeated: Echocardiography, clinical evaluation, pacemaker test and blood samples. Rb-PET is also repeated to determine potential changes in myocardial perfusion and LVEF. Thereafter the patient will attend standard controls of the pacemaker every six month according to standard procedures.

Power Calculations and statistics:

We hypothesize that a CRT-strategy targeting optimal electrical resynchronization will result in an excess increase of 4 % in LVEF compared with the routine CRT-strategy, where an 8 % increase is expected. To identify this absolute increase in LVEF and to achieve a statistical power of 80 %, the study will need a sample size of 98 patients, given a standard deviation (SD) of 7 % in both groups, and a two-sided alpha value of 0.05. Furthermore, to achieve a statistical power of > 80 % with a margen of noninferiority of 20 % for the secondary endpoint of clinical non-response to CRT (assuming a 75 % clinical response rate in the control group) we will need a sample size of 116 patients (given a two-sided alpha value of 0.05 %). Taking into consideration an expected loss of follow-up in approximately 5 % of the patients, we will include 122 patients.

All analyses will be conducted according to the intention-to-treat principle. Differences between groups will be tested using Students t-test, when normality is demonstrated; otherwise a non-parametric test (Mann-Whitney) is used. Categorical variables will be analyzed by χ2 test. A two-sided P- value of <0.05 is considered significant.

Research Plan:

The Department of Cardiology, Aarhus University Hospital, have the capacity and equipment to conduct this trial. The group of investigators contributes with a deep and long-lasting experience in CRT-treatment and 150 de-novo CRT-devices are annually implanted at our institution. We plan to enroll the patients during a two and a half-year period. This study is planned to start in February 2015 as a PhD program for Charlotte Stephansen, MD. Charlotte Stephansen will be the prime investigator in charge of including the patients and she will perform all clinical evaluations and image acquisitions during the admission for CRT implantation and at the six month follow-up. She will also be in charge of analyzing data after study completion.

The results will be published in peer-reviewed international journals, and are expected to result in at least three papers. None of the investigators have any conflicts of interest to declare.

The study will be conducted according to the principles of the Helsinki Declaration II. The study will be approved by The Central Denmark Region Committees on Health Research Ethics, reported to the Danish Data Protection Agency, and registered on ClinicalTrials.gov.

Perspective:

No prospective randomized trials have previously investigated the effect of a CRT treatment-strategy targeting optimal electrical resynchronization achieved by guiding LV lead placement to the myocardial region with the latest electrical activation combined with post-implant VV electrical optimization for narrowing the paced QRS width.

It is expected that this method improves the response to CRT. The human and economic costs of CRT in non-responders are therefore expected to be reduced. If an excess increase in LVEF is achieved in this study, it will be possible to prevent and relieve invalidating symptoms and reduce mortality in selected heart failue patients in the future. The utility and potential benefits of participating in this study are expected to equalize the risks of exposure to ionizing radiation, possible side effects and inconvenience to the patient.

References:

Please refer to the reference chapter

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure (New York Heart Association (NYHA) functional class II - IV) despite optimal medical therapy
* ECG with left bundle branch block and QRS ≥ 120 ms
* LVEF ≤ 35 %
* Age > 40 years
* Written informed consent Patients with an indwelling single- or dual chamber pacemaker and a paced QRS > 180 ms are eligible for enrollment.

Exclusion Criteria:

* Expected lifetime < 6 months
* Expected heart-surgery within the next 6 months
* Recent (< 3 months) myocardial infarction or coronary artery bypass graft (CABG)
* Pregnant or lactating
* No written informed consent Cardiac CT will not be performed in patients where this is contraindicated, i.e. in the presence of depressed renal function (estimated Glomerular Filtration Rate (eGFR) < 30 ml (milliters)/minute), thyrotoxicosis or in the case of former serious reactions to the contrast media.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | The day before implantation and 6 months after implantation
  Change in LVEF determined by 2D echocardiography

SECONDARY OUTCOMES:
All cause mortality | 6 months and until "3 years and 6 months" after implantation
  The patients will be asked to give permission to pass along information from their cardiovascular medical records to the primary investigator until three years after the six months follow-up evaluation
Hospitalization for heart failure | 6 months and until "3 years and 6 months" after implantation
  The patients will be asked to give permission to pass along information from their cardiovascular medical records to the primary investigator until three years after the six months follow-up evaluation
CRT-implant procedure time | The day of implantation
  During implatation procedure
Procedural radiation exposure | The day of implantation
  During implantation procedure
Perioperative and late complications | The day of implantation, 6 months and until "3 years and 6 months" after implantation
  Procedural and retrospective. The patients will be asked to give permission to pass along information from their cardiovascular medical records to the primary investigator until three years after the six months follow-up evaluation
Changes in Quality of Life | The day before implantation and 6 months
  Changes in Quality of Life Assessed by Minnesota Living With Heart Failure Questionnaire
Changes in New York Heart Association Functional Class | The day before implantation and 6 months
  Changes in New York Heart Association Functional Class assesed by clinical evaluation
Changes in Six Minutes Walk Test | The day before implantation and 6 months
Changes in level of N-terminal prohormone of brain natriuretic peptide | The day before implantation and 6 months
  Changes in level of N-terminal prohormone of brain natriuretic peptide blood sample
Changes in Left Ventricular End Systolic Volume | The day before implantation and 6 months
  Changes in Left Ventricular End Systolic Volume assessed by 2D echocardiography and Rb-PET
Changes in Left Ventricular End Diastolic Volume | The day before implantation and 6 months
  Changes in Left Ventricular End Diastolic Volume assessed by 2D echocardiography and Rb-PET
Changes in Electrode Parameters (pacing threshold, sensing value, impedance) | The day after implantation and at 1 and 6 months follow-up
  Changes in Electrode Parameters (pacing threshold, sensing value, impedance) assessed by pacemakertest
Changes in Echocardiographic Dyssynchrony parameters | The day before implantation and at 6 months follow-up
  Determined by 2D echocardiography
Clinical response to CRT at 6 months follow-up if the patient is: 1. Alive, and 2. Not hospitalized for heart failure, and 3. experience an improvement of NYHA Functional Class or > 10 % increase in 6MWT | At the 6 months follow-up.
  The patients will be asked to give permission to pass along information from their cardiovascular medical records to the primary investigator until three years after the six months follow-up evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jens Cosedis Nielsen, Professor, Study Director — Aarhus University Hospital, Sekjby, Department of Cardiology; Mads Brix Kronborg, MD, PhD, Study Director — Aarhus University Hospital, Sekjby, Department of Cardiology; Anders Sommer Knudsen, MD, Study Director — Aarhus University Hospital, Sekjby, Department of Cardiology
Locations (1):
- Aarhus University Hospital, Skejby, Department of Cardiology, Aarhus, Denmark

REFERENCES:
- [Background] European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE. 2013 ESC guidelines on cardiac pacing and cardiac resynchronization therapy: the task force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Europace. 2013 Aug;15(8):1070-118. doi: 10.1093/europace/eut206. Epub 2013 Jun 24. No abstract available. PMID 23801827
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Yu CM, Sanderson JE, Gorcsan J 3rd. Echocardiography, dyssynchrony, and the response to cardiac resynchronization therapy. Eur Heart J. 2010 Oct;31(19):2326-37. doi: 10.1093/eurheartj/ehq263. Epub 2010 Aug 13. PMID 20709721
- [Background] Kronborg MB, Mortensen PT, Kirkfeldt RE, Nielsen JC. Very long term follow-up of cardiac resynchronization therapy: clinical outcome and predictors of mortality. Eur J Heart Fail. 2008 Aug;10(8):796-801. doi: 10.1016/j.ejheart.2008.06.013. Epub 2008 Jul 10. PMID 18619900
- [Background] Kirkfeldt RE, Johansen JB, Nohr EA, Jorgensen OD, Nielsen JC. Complications after cardiac implantable electronic device implantations: an analysis of a complete, nationwide cohort in Denmark. Eur Heart J. 2014 May;35(18):1186-94. doi: 10.1093/eurheartj/eht511. Epub 2013 Dec 17. PMID 24347317
- [Background] Gold MR, Birgersdotter-Green U, Singh JP, Ellenbogen KA, Yu Y, Meyer TE, Seth M, Tchou PJ. The relationship between ventricular electrical delay and left ventricular remodelling with cardiac resynchronization therapy. Eur Heart J. 2011 Oct;32(20):2516-24. doi: 10.1093/eurheartj/ehr329. Epub 2011 Aug 29. PMID 21875862
- [Background] Kandala J, Upadhyay GA, Altman RK, Parks KA, Orencole M, Mela T, Kevin Heist E, Singh JP. QRS morphology, left ventricular lead location, and clinical outcome in patients receiving cardiac resynchronization therapy. Eur Heart J. 2013 Aug;34(29):2252-62. doi: 10.1093/eurheartj/eht123. Epub 2013 Apr 9. PMID 23571836
- [Background] Kronborg MB, Nielsen JC, Mortensen PT. Electrocardiographic patterns and long-term clinical outcome in cardiac resynchronization therapy. Europace. 2010 Feb;12(2):216-22. doi: 10.1093/europace/eup364. Epub 2009 Nov 14. PMID 19915182
- [Background] Tamborero D, Vidal B, Tolosana JM, Sitges M, Berruezo A, Silva E, Castel M, Matas M, Arbelo E, Rios J, Villacastin J, Brugada J, Mont L. Electrocardiographic versus echocardiographic optimization of the interventricular pacing delay in patients undergoing cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2011 Oct;22(10):1129-34. doi: 10.1111/j.1540-8167.2011.02085.x. Epub 2011 Jun 2. PMID 21635609
- [Background] Tamborero D, Mont L, Sitges M, Silva E, Berruezo A, Vidal B, Delgado V, Tolosana JM, Godoy M, Castel A, Brugada J. Optimization of the interventricular delay in cardiac resynchronization therapy using the QRS width. Am J Cardiol. 2009 Nov 15;104(10):1407-12. doi: 10.1016/j.amjcard.2009.07.006. PMID 19892059
- [Background] Ypenburg C, Schalij MJ, Bleeker GB, Steendijk P, Boersma E, Dibbets-Schneider P, Stokkel MP, van der Wall EE, Bax JJ. Impact of viability and scar tissue on response to cardiac resynchronization therapy in ischaemic heart failure patients. Eur Heart J. 2007 Jan;28(1):33-41. doi: 10.1093/eurheartj/ehl379. Epub 2006 Nov 22. PMID 17121757
- [Background] Bravo PE, Chien D, Javadi M, Merrill J, Bengel FM. Reference ranges for LVEF and LV volumes from electrocardiographically gated 82Rb cardiac PET/CT using commercially available software. J Nucl Med. 2010 Jun;51(6):898-905. doi: 10.2967/jnumed.109.073858. Epub 2010 May 19. PMID 20484424
- [Background] Sommer A, Kronborg MB, Norgaard BL, Gerdes C, Mortensen PT, Nielsen JC. Left and right ventricular lead positions are imprecisely determined by fluoroscopy in cardiac resynchronization therapy: a comparison with cardiac computed tomography. Europace. 2014 Sep;16(9):1334-41. doi: 10.1093/europace/euu056. Epub 2014 Mar 30. PMID 24687965
- [Derived] Stephansen C, Sommer A, Kronborg MB, Jensen JM, Bouchelouche K, Nielsen JC. Electrically guided versus imaging-guided implant of the left ventricular lead in cardiac resynchronization therapy: a study protocol for a double-blinded randomized controlled clinical trial (ElectroCRT). Trials. 2018 Nov 1;19(1):600. doi: 10.1186/s13063-018-2930-y. PMID 30382923